CLINICAL TRIAL: NCT04500834
Title: Clinical Evaluation of Metal Panel Allergens: Safety and Efficacy Study
Brief Title: Metal Panel Allergen Patch Test Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SP20 11MP 301
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Intervention Model Description: All subjects will be tested with 11 experimental metal allergens and corresponding metal allergens prepared in petrolatum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Positive reactions, Concordance with reference allergen (Experimental): All subjects will be patch tested with 11 experimental and 11 reference allergens. Rates of positive reactions will be evaluated using Cohen's kappa calculation.
  Interventions: Biological: Metal Panel T.R.U.E. Test

INTERVENTIONS:
Biological: Metal Panel T.R.U.E. Test — Diagnostic patch test

SUMMARY:
Metal allergen patch test study.

DETAILED DESCRIPTION:
A single application of an investigational patch test panel containing 11 hydrogel metal allergens and a corresponding patch test panel containing 11 petrolatum metal allergens will be applied to the upper back of human subjects to test diagnostic efficacy and safety. Patch test panels will be removed after being worn for approximately 48 hours. Study will require 6 visits over the course of 21 days; patch application, patch removal and 4 patch test site evaluation visits at days 4, 7, 14 and 21.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Past positive patch test result within the past 10 years to one of the metal allergens (other than nickel or gold), being tested on this study or strong suspicion of metal contact allergy based on results of the Qualification Questionnaire, part 2 Type of Metal Exposure.
3. Unable to become pregnant or willing to use an acceptable method of contraception to prevent pregnancy if female of childbearing potential,

   * Inability to become pregnant would include all male subjects and female subjects who are postmenopausal for at least 1 year, or surgically sterile- have had a hysterectomy, bilateral ovariectomy, uterine ablation or bilateral tubal ligation.
   * Acceptable methods of contraception include: 1) systemic birth control (i.e., oral contraceptives, skin patch, vaginal ring, implant, injection, or intrauterine device (IUD), which contains either a hormone or copper); 2) double barrier method (i.e., diaphragm, cervical cap, sponge, condom with spermicide); 3) IUD; 4) vasectomized partner; or 5) abstinence from sexual intercourse. Subject must agree to use acceptable contraception for the duration of the entire study.
4. Understands and signs the approved Informed Consent form which is consistent with all institutional, local and national regulations.

Exclusion Criteria:

1. Breastfeeding or pregnant (as determined by urine pregnancy test) or intending to become pregnant during the course of the study. Breastfeeding may be resumed upon completion of the study.
2. Topical treatment with corticosteroids or other immunosuppressive agents on or near the test area 14 days prior to inclusion through the end of the subject's participation in the study.
3. Systemic treatment with corticosteroids (equivalent to > 10 mg prednisone) or other immunosuppressive agents 14 days prior to inclusion through the end of the subject's participation in the study. Inhaled treatments and steroidal nose or eye drops are permitted.
4. Treatment with ultraviolet (UV) light (including tanning) during the 3 weeks prior to inclusion through the end of the subject's participation in the study.
5. Acute dermatitis outbreak or dermatitis on or near the test area on the back.
6. Known or suspected infection of the skin, joints or other site(s) associated with metal exposure
7. Condition such as; fibromyalgia, chronic fatigue, depression, cognitive impairment, flu-like symptoms, diarrhea and/or headache without at least one of the symptoms related to metal exposure listed in Section 6.6.
8. Condition such as; psoriasis, dermatitis herpetiformis, mycosis fungoides or cutaneous T-cell lymphoma that may confound the evaluation of allergic contact dermatitis.
9. Inability to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).
10. Participation in a clinical trial of an investigational drug, treatment or device during this study or 3 weeks prior to inclusion in this study.
11. An opinion of the Investigator that deems the potential subject to be non-compliant, unable to return for study visits or complete the study as detailed in the protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with positive, negative, irritant or doubtful patch test responses and concordance between hydrogel and petrolatum allergens | Days 3-21
  Number of patch test responses will be recorded, concordance between hydrogel and petrolatum allergens will be measured

SECONDARY OUTCOMES:
Evaluation of panel adhesion at visit 2 prior to panel removal | Day 2
  Number of subjects with excellent, good, poor or detached adhesion at panel removal
Evaluation of subject reported itching associated with test panels at visit 2 following panel removal | Day 2
  Number of subjects with no (none) weak, moderate or strong itching associated with test panels following panel removal
Evaluation of subject reported burning associated with test panels at visit 2 following panel removal. | Day 2
  Number of subjects with no (none) weak, moderate or strong burning associated with test panels following panel removal
Evaluation of tape irritation | Day 21
  Number of subjects with no (none) irritant or allergic tape irritation. Tape irritation is assessed at all visits. Investigator makes overall determination on day 21.
Evaluation of chip irritation | Day 21
  Number of subjects with no (none) irritant or allergic chip irritation. Chip irritation is assessed at all visits. Investigator makes overall determination on day 21.

CONTACTS AND LOCATIONS:
Overall Officials: Curt Hamann, M.D., Study Director — Allerderm (dba SmartPractice)
Locations (1):
- DS Research, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.